CLINICAL TRIAL: NCT04063254
Title: A Prospective Randomized Trial of High Dose Versus Standard Dose Stereotactic Radiotherapy for Pain Control in Patients With Bone Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201906063RINB
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Bone Metastases; Radiotherapy Side Effect
MeSH Terms: conditions — Radiation Injuries | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dose Stereotactic Radiotherapy (Experimental)
  Interventions: Radiation: Stereotactic Radiotherapy
- Standard-Dose Stereotactic Radiotherapy (Active Comparator)
  Interventions: Radiation: Stereotactic Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Radiotherapy — High Dose (Arm A): Stereotactic radiotherapy with 12 or 16 Gy in single fraction using intensity modulated radiotherapy or volumetric modulated arc therapy (VMAT or RapidArc).
  Standard-dose (Arm B): Stereotactic radiotherapy with 8 or 10 Gy in single fraction using intensity modulated radiotherapy or volumetric modulated arc therapy (VMAT or RapidArc).

SUMMARY:
In the present study, we will prospectively evaluate the pain response and treatment failure rate to determine the most favorable radiation dose in single fraction stereotactic radiotherapy using the modern highly conformal technique for bone metastases. Our findings should be able to provide evidence-based recommendation to support the utilization of single fraction radiotherapy for value-based oncology practice.

DETAILED DESCRIPTION:
Primary objective To evaluate dose regimen for pain control in terms of rate of treatment failure, defined as the first occurrence of any of the following events, at 3 months

1. Worsening in the worst pain score by at least 3 by brief pain inventory survey
2. ≥ 50% increase in dose of opioid/narcotic medication
3. Development of pathologic fracture or cord/nerve compression indicative of surgical intervention
4. Unequivocal radiographic disease progression

Secondary objectives

1. Compare pain response/control at the treated site(s) between the two treatment regimens by brief pain inventory survey
2. Assess health-related quality of life for palliative cancer care patients (EORTC QLQ-C15-PAL & EORTC-BM22 Mandarin Taiwan)
3. Evaluate the analgescis use after irradiation
4. Evaluate acute and late adverse events associated with irradiation according to CTCAE criteria
5. To evaluate the local control of the treated index site(s)
6. To evaluate the patterns of failure
7. To evlaute overall survival
8. To evaluate the rate of re-irradiation, salvage surgery, interventional procedure, and MR-guided high intensity focused ultrasound at the treated site(s)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologic diagnosis of non-hematopoietic malignancy
2. Radiographic evidence of bone metastases
3. Patient with pain or dysathesia on a pain score of at least 2 by brief pain inventory survey
4. Multiple osseous sites are eligible with a maximum of three separate sites irradiated concurrently
5. Patients do not have prior radiotherapy or radiosurgery to the index site(s)
6. Age ≥ 20 years
7. Karnofsky performance status (KPS) ≥ 50%.
8. Life expectancy of ≥ 3 months
9. Women of childbearing potential and male participants must practice adequate contraception
10. Patients must be able to comply with the study protocol, pain assessment, quality of life survey, and follow-up schedules and provide study-specific informed consent

Exclusion Criteria:

1. Patients with radiographic impending or pathological fracture, or malignant epidural cord compression at the index site(s) indicative of upfront surgery
2. Prior radiotherapy or radiosurgery to the index site(s)
3. Previously treated with radioactive isotope (e.g. Ra-223) within 30 days of registration
4. Inability to cooperate treatment procedure
5. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

   1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
   2. Transmural myocardial infarction ≤ 6 months prior to registration
   3. Unstable angina or congestive heart failure requiring hospitalization ≤ 6 months prior to registration
   4. Life-threatening uncontrolled clinically significant cardiac arrhythmias
   5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   6. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   7. Uncontrolled psychiatric disorder
6. Will receive any other investigational agent or chemotherapy during treatment
7. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic
8. Pregnant or breast-feeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Effects of treatment | 3 months
  To evaluate dose regimen for pain control in terms of rate of treatment failure, defined as the first occurrence of any of the following events

IPD SHARING:
Plan to Share IPD: Undecided